CLINICAL TRIAL: NCT00420602
Title: Clinical Interventions Against Stargardt Macular Dystrophy: DHA Supplementation in Patients With STGD3
Brief Title: DHA Supplementation in Patients With STGD3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Paul S. Bernstein, Professor of Ophthalmology, University of Utah
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IRB 19676
Record Dates: First submitted 2007-01-10; First posted 2007-01-11 (Estimated); Last update posted 2018-05-09 (Actual); Status verified 2018-05

CONDITIONS: Dominantly Inherited Stargardt's Disease (STGD3)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single Arm, Open Label (Other): Single Arm, Open Label
  Interventions: Dietary Supplement: Over the counter DHA/EPA dietary supplementation

INTERVENTIONS:
Dietary Supplement: Over the counter DHA/EPA dietary supplementation — 1000 mg/day DHA/EPA

SUMMARY:
We have found that biomarkers of long-term elevated dietary intake of omega-3 fatty acids such as DHA and EPA are inversely associated with severity of disease phenotype in STGD3 patients. Therefore, the purpose of this study is to follow STGD3 patients as they supplement their diets with DHA/EPA.

ELIGIBILITY:
Inclusion Criteria:

* All Moran Eye Center patients with STGD3

Exclusion Criteria:

* All others

Ages: 18 Years to 105 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2007-09-21 (Actual); Primary Completion 2017-12-27 (Actual); Study Completion 2017-12-27 (Actual)

PRIMARY OUTCOMES:
ERG | 1 year

SECONDARY OUTCOMES:
Visual acuity | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Paul S. Bernstein, MD Ph.D., Principal Investigator — University of Utah
Locations (1):
- Moran Eye Center, University of Utah, Salt Lake City, Utah, United States